CLINICAL TRIAL: NCT00320879
Title: Optimal Dose of Irbesartan for Renoprotection in Type 2 Diabetic Patients With Persistent Microalbuminuria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 26122284
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2006-05-18 (Estimated); Status verified 2003-07

CONDITIONS: Type 2 Diabetes; Microalbuminuria
Keywords: diabetes; microalbuminuria; angiotensin II receptor blockade; irbesartan; dose-response; randomized; double-blind; renin-angiotensin-aldosterone system; clinical; hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hypertension | interventions — Irbesartan

INTERVENTIONS:
Drug: irbesartan

SUMMARY:
Aim: To evaluate the renoprotective effect as reflected by short-term changes in albuminuria of ultra high doses of irbesartan in Type 2 diabetic patients with microalbuminuria Design: A double-masked randomized cross-over trial including 60 hypertensive Type 2 diabetic patients with microalbuminuria on ongoing antihypertensive medication. At inclusion, previous antihypertensive treatment will be discontinued and replaced with bendroflumethiazide 5 mg o.d. for the entire study. Following two months wash-out (baseline), patients will be treated randomly with irbesartan 300, 600 and 900 mg o.d., each dose for two months. End-points evaluated at the end of each study period include urinary albumin excretion rate (UAE, mean of three 24-hrs collections), 24-hrs blood pressure (ABP); and GFR (51Cr-EDTA).

DETAILED DESCRIPTION:
Aim:

The primary aim of our study is to evaluate the antiproteinuric effect of irbesartan 300, 600 and 900 mg once daily in type 2 diabetic patients with microalbuminuria. Secondary to evaluate the effect on 24-h ambulatory blood pressure, glomerular filtration rate (GFR), urinary TGF beta excretion, and markers of endothelial dysfunction, and finally to evaluate the association between treatment response and genotypes with possible implications for the risk of cardiovascular disease.

Patients 60 type 2 diabetic patients with persistent microalbuminuria (at least two out of three 24-h urinary collections with albumin excretion between 30 and 300 mg/24-h).

Duration of study 38 weeks (8 weeks wash-out and 30 weeks of double-blind randomized cross-over (treatment with irbesartan 300, 600 and 900 mg for 10 weeks at each dose level)).

Design The study consists of an eight week wash-out period followed by a double-blind randomized three 10 week treatment period cross-over trial (please see enclosed flow chart).

Wash-out period: Eight weeks prior to randomization all previous antihypertensive medication is discontinued and replaced by hydrochlorothiazide 25 mg once daily throughout the entire study period. Hydrochlorothiazide is added to reduce blood pressure elevation and edema formation during the trial and to eliminate the influence of varying dietary salt intake on the effects of irbesartan during the double blind treatment periods.

Double-blind cross-over periods: All patients receive treatment with irbesartan 300, 600 and 900 mg once daily in random order, without wash-out between treatment periods. All treatment periods are of 10 weeks duration. They consist of an initial two week titration period on irbesartan 300 mg o.d. to minimize the risk of adverse events including hypotension during cross-over in doses followed by an eight week period on the full dose for the given treatment level.

For safety reasons blood pressure, serum potassium and serum creatinine will be measured 4 weeks after the beginning of each treatment period (two weeks after the full dose of the treatment period is reached).

End-points are evaluated after the wash-out period (baseline) and at the end of each treatment period.

Methods Albuminuria is assessed by turbidimetry in three 24-h urinary samples. 24-h ambulatory blood pressure by the Takeda TM-2420/2421 device. GFR by plasma clearance of 51Cr-EDTA. DNA will be extracted from a venous sample to determine genotypes with possible implications for the risk of cardiovascular disease. Initially we will evaluate the influence of the ACE/ID- , Angiotensin II type I receptor (A1166C) - and the angiotensinogen (M235T) polymorphisms.

Endpoints Primary endpoint: change in albuminuria Secondary endpoints: 24-h ambulatory blood pressure, glomerular filtration rate (GFR), and to evaluate the association between treatment response genotypes with possible implications for the risk of cardiovascular disease

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (WHO criteria) and age above 18 years.
* Persistent microalbuminuria (urinary albumin excretion between 30 and 300 mg/24-h in at least two out of three 24-urinary collections
* Systolic blood pressure > 110 mmHg

Exclusion Criteria:

* Serum creatinine > 150 micromol/l
* Known non-diabetic renal disease
* Pregnancy or fertile women not using adequate contraception (intrauterine device, sterilization or oral anticonception)
* Systolic blood pressure persistently > 180 mm Hg or < 100 mm Hg
* Diastolic blood pressure persistently > 105 mm Hg
* Plasma potassium > 4.8 mmol/l
* Heart failure, acute myocardial infarction, unstable angina or coronary by-pass surgery within the previous three months.
* Known intolerance to angiotensin II receptor blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52
Dates: Start 2003-09; Study Completion 2004-11

PRIMARY OUTCOMES:
urinary albumin excretion rate

SECONDARY OUTCOMES:
ambulatory blood pressure
glomerular filtration rate
serum potassium
serum creatinine
lipids
renin
aldosterone
NT-proBNP
markers of endothelial function
markers of inflammation
genotypes with possible implications for the risk of cardiovascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Henrik Parving, Study Director — Steno Diabetes Center, Gentofte, Denmark; Kasper Rossing, Principal Investigator — Steno Diabetes Center, Gentofte, Denmark
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Copenhagen, Denmark

REFERENCES:
- [Result] Rossing K, Schjoedt KJ, Jensen BR, Boomsma F, Parving HH. Enhanced renoprotective effects of ultrahigh doses of irbesartan in patients with type 2 diabetes and microalbuminuria. Kidney Int. 2005 Sep;68(3):1190-8. doi: 10.1111/j.1523-1755.2005.00511.x. PMID 16105050